CLINICAL TRIAL: NCT06796868
Title: A Multicenter, Randomized , Double-blind, Parallel, Placebo-controlled Design Clinical Trial of GW117 Tablets
Brief Title: A Study to Evaluate Efficacy and Safety of GW117 Tablets in Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Greatway Pharmaceutical Technology Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GW117-C201
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — GW117

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- GW117 Tablets 20mg group (Experimental)
  Interventions: Drug: GW117 Tablets
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- GW117 Tablets 40mg group (Experimental)
  Interventions: Drug: GW117 Tablets
- GW117 Tablets 60mg group (Experimental)
  Interventions: Drug: GW117 Tablets

INTERVENTIONS:
Drug: GW117 Tablets — GW117 Tablets 20mg orally once a day
  Arms: GW117 Tablets 20mg group
Drug: GW117 Tablets — GW117 Tablets 20mg*2 orally once a day
  Arms: GW117 Tablets 40mg group
Drug: GW117 Tablets — GW117 Tablets 20mg*3 orally once a day
  Arms: GW117 Tablets 60mg group
Drug: Placebo — placebo orally once a day
  Arms: placebo

SUMMARY:
The study aims to evaluate the efficacy and safety of GW117 Tablets compared to placebo in adults participants with MDD over a period of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 18 to 65 years (including both limits), either male or female;
* Meet the diagnostic criteria for depression in DSM-5 (the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders), without psychotic symptoms;
* Have a total score of ≥ 22 on the 17-item Hamilton Depression Rating Scale (HAM-D17) at both screening and baseline visits;
* Have a Clinical Global Impression - Severity (CGI-S) score of ≥ 4 at both screening and baseline visits;
* Voluntarily participate in this trial and sign the informed consent form, and be able to comply with the planned visits, treatment plan, laboratory tests and other research procedures.

Exclusion Criteria:

* Allergic constitution (such as those allergic to two or more drugs or foods) or known to be allergic to similar products like agomelatine;
* Have previously received adequate and full-course treatment with agomelatine but showed no effect, or treatment-resistant depression (those who have used at least two antidepressants in adequate and full-course treatment but still showed no effect);
* HAM-D17 scale score reduction rate is ≥25% compared to the baseline period;
* High suicide risk; history of suicide attempts within one year before screening; suicidal or self-harming behavior during the screening period; score of ≥3 on item 3 (suicide item) of the HAM-D17 scale;
* Diagnosed with any disease other than depression according to DSM-5, including anxiety disorders, neurodevelopmental disorders, schizophrenia spectrum and other psychotic disorders, bipolar and related disorders, obsessive-compulsive and related disorders, trauma and stress-related disorders, dissociative disorders, anorexia or bulimia nervosa, personality disorders, etc.;
* Depression secondary to other mental or physical diseases. Note: Other inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
The change in Hamilton Depression Scale-17(HAMD-17) total score from baseline | 8 week
  There are a total of 17 projects in Hamilton Depression Scale-17（HAMD-17）. Scores are distributed on a scale of 0 to 53. Higher scores represent a more severe condition.

SECONDARY OUTCOMES:
The change inMontgomery-Åsberg Depression Rating Scale (MADRS) total score from baseline | 8 week
  There are a total of 10 projects in Montgomery-Asberg Depression Rating Scale（MADRS）, each with a 7-point scoring system ranging from 0 to 6 points,for a total possible score of 60. The higher the score, the more severe the degree of depression.
The response rate of HAMD-17 | 8 week
  The response definition of HAMD-17 is that the reduction rate of HAMD-17 score relative to baseline is ≥ 50%.
The response rate of MADRS | 8 week
  The response definition of MADRS is that the reduction rate of MADRS score relative to baseline is ≥ 50%.
The changes in Clinical Global Impression Scale-Improvement (CGI-I )total score from baseline | 8 week
  the following one query is rated on a seven-point scale: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment. the higher the score, the more severe the condition will be.
The changes in Clinical Globel Impression-Severity(CGI-S) from baseline | 8 week
  The CGI-Severity (CGI-S) is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
  This rating is based upon observed and reported symptoms, behavior, and function in the past seven days. the score should reflect the average severity level across the seven days.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Hebei Mental Health Center, Baoding
  - Beijing Huilongguan Hospital, Beijing
  - Capital Medical University Affliated Anding HospitalContact, Beijing
  - Peking University Sixth Hospital, Beijing
  - Chengdu No.4 People's Hospital, Chengdu
  - Chongqing Mental Health Center, Chongqing
  - The third hospital of Daqing, Daqing
  - Huzhou Third People's Hospital, Huzhou
  - Jilin Neuropsychiatric Hospital, Jilin
  - The Third People's Hospital of Mianyang City, Mianyang
  - Shanghai Mental Health Center, Shanghai
  - Shenzhen Kangning Hospital, Shenzhen
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Anding Hospital, Tianjin
  - Wuxi Mental Health Center, Wuxi
  - Xijing Hospital, the Fourth Military Medical University, Xi'an, China, Xi'an
  - Zhumadian Second People's Hospital, Zhumadian

REFERENCES:
- [Derived] Shen Y, Hao X, Shi X, Tao Z, Yu X, Wang X, Di X, Yang H, Zhang Y, Li J, Wang Z, Zhang G, Wang J, Jiang Z, Wang R, Liu J, Dong Z, Gu W, Zhang H. Efficacy and safety of GW117 tablets in major depressive disorder: a randomised, double-blind, placebo-controlled, phase 2 dose-finding study. Gen Psychiatr. 2025 Dec 17;38(6):e102337. doi: 10.1136/gpsych-2025-102337. eCollection 2025. PMID 41425080